CLINICAL TRIAL: NCT02415504
Title: Comprehensive Care Transition: A Randomized Control Trial of an Enhanced Care Transition Process in Dementia
Brief Title: Comprehensive Care Transition: A Trial of an Enhanced Care Transition Process in Dementia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding problems, slow recruitment, PI location change
Sponsor: Baycrest (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Dr. Colleen Ray, Ph.D., C.Psych, Baycrest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB14-45
Record Dates: First submitted 2014-12-05; First posted 2015-04-14 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Dementia; BPSD
Keywords: Care transition; Behavioural and psychological symptoms of dementia; BPSD; Dementia; Persons with dementia; Discharge processes
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced care transition (Experimental): The enhanced care transition will offer: (1) an integrated behavioural care plan, (2) an in- person discharge meeting including family, post-care transition staff (LTC or another hospital unit) and unit staff, (3) videos of responsive behaviours and non-pharmacological interventions, (4) a briefcase of favoured activities, (5) an in-person care demonstration, and (6) involvement of a transitional care team.
  Interventions: Behavioral: Enhanced care transition
- Standard care transition (Other): The standard care transition varies by unit, and either consists of: (1) a discipline specific care plan, (2) a phone discharge meeting between unit staff and post-care transition staff (LTC or another hospital unit) and (3) a follow-up phone call with social work OR (1) a discipline specific care plan, (2) an in-person meeting between unit staff and (family) caregivers, (3) involvement of a transitional care team, and (4) a follow-up phone call with social work.
  Interventions: Behavioral: Standard care transition

INTERVENTIONS:
Behavioral: Enhanced care transition — Enhanced care transition discharge package: (1) an integrated behavioural care plan, (2) an in-person discharge meeting including family, post-care transition staff (LTC or another hospital unit) and unit staff, (3) videos of responsive behaviours and non-pharmacological interventions, (4) a briefcase of favoured activities, (5) an in-person care demonstration, and (6) involvement of a transitional care team.
  Arms: Enhanced care transition
Behavioral: Standard care transition — Standard care transition discharge package: The standard care transition varies by unit, and either consists of: (1) a discipline specific care plan, (2) a phone discharge meeting between unit staff and post-care transition staff (LTC or another hospital unit) and (3) a follow-up phone call with social work OR (1) a discipline specific care plan, (2) an in-person meeting between unit staff and (family) caregivers, (3) involvement of a transitional care team, and (4) a follow-up phone call with social work.
  Arms: Standard care transition

SUMMARY:
This pilot study examines the impact of an enhanced care transition process vs. usual care for persons with dementia admitted to a transitional unit (hospital or LTC) for management of behavioural and psychological symptoms of dementia (BPSD) with a planned discharge to long term care (LTC) facilities or other hospital units. Deficiencies in discharge processes can contribute to poor outcomes (e.g., readmissions), and there is a dearth of research on how to improve care transitions for persons with BPSD. The investigators aim to improve the care transition process for persons with dementia and BPSD utilizing an enhanced care transition process that will contain up to 6 elements: integrated behavioural care plans, videos, patient specific briefcase containing activities to reduce BPSD, in-person care transition meeting, in-person care demonstration (when possible), and follow up visits with a transition team. The ability to determine the effect of enhanced care transitions on the clinical course of patients with planned discharge to LTC or hospital may allow for improved outcomes and an overall increased efficiency of post discharge care.

DETAILED DESCRIPTION:
The investigators have formulated an enhanced care transition process based on factors that have been documented to support care transitions in other clinical populations (e.g., Coleman, 2003 on persons with continuous complex needs; Viggiano, et al., 2012 on persons with mental health issues), along with novel package elements based on the investigators' experience working with persons with dementia and BPSD. The investigators propose to conduct a preliminary analysis of patient and staff outcomes comparing an enhanced care transition process with a control group receiving usual care. The investigators' proposed enhanced care transition process will contain 5 elements: 1. Unified transfer care document adapted to the post-care transition location 2. Videos of BPSD management to better communicate care provision, 3. Provision to -the post-care transition location a patient specific briefcase containing activities that help to reduce BPSD, 4. In-person care transition meeting between sites, including the family, to transfer knowledge, 5. In person care demonstration (when possible), and 6. Follow-up visits post transition with a transition team (a service already in existence but not consistently used). The investigators hope that with improved communication, discharge locations will be better equipped to manage BPSD, and reduce the likelihood of adverse events for both patients and staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients on behavioural transitional support unit's at Baycrest (Behavioural Neurology Unit, transitional Behavioural Support Unit) who are admitted for behavioural and psychological symptoms of dementia (BPSD)
* Diagnosed with a degenerative dementia
* Over 55 years old at the time of discharge, with a planned discharge to a long-term care (LTC) facility or another hospital unit will be eligible for the study

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Post-Care Transition (PCT) questionnaire | Change in resident's baseline behaviour(s) at 2 and 4 weeks
  Likert scales and open-ended questions measuring change in the transitioned resident's identified behaviour(s).

SECONDARY OUTCOMES:
Social work assessment questionnaire | At 6 months after baseline
  Likert scales and open-ended questions evaluating the transition process and the post-care transition location.
Substitute Decision Maker (SDM) satisfaction questionnaire | At baseline
  Likert scales and open-ended questions measuring the SDM's satisfaction with resident's transition.
Substitute Decision Maker (SDM) satisfaction questionnaire | Change from baseline at 2 weeks
  Likert scales and open-ended questions measuring the SDM's satisfaction with resident's transition.
Substitute Decision Maker (SDM) questionnaire | At baseline
  Likert scales and open-ended questions measuring the SDM's perception of the resident's identified baseline behaviour(s).
Substitute Decision Maker (SDM) questionnaire | Change in resident's baseline behaviour(s) at 2 and 4 weeks
  Likert scales and open-ended questions measuring the SDM's perception of change in the transitioned resident's identified behaviour(s).
Post-Care Transition (PCT) questionnaire | Change in resident's baseline behaviour(s) at 3 and 6 months
  Likert scales and open-ended questions measuring change in the transitioned resident's identified behaviour(s).
Post-Care Transition (PCT) staff satisfaction questionnaire | Change from baseline at 2 and 4 weeks
  Likert scales and open-ended questions evaluating staff satisfaction with the resident's transition process.
Chart review | At baseline
  Resident's additional dependent data collection (e.g., demographics, identified behaviours, Cohen Mansfield Agitation Inventory score, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Ray, PhD, Principal Investigator — Neuropsychology and Cognitive Health at Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viggiano T, Pincus HA, Crystal S. Care transition interventions in mental health. Curr Opin Psychiatry. 2012 Nov;25(6):551-8. doi: 10.1097/YCO.0b013e328358df75. PMID 22992544
- [Background] Coleman EA. Falling through the cracks: challenges and opportunities for improving transitional care for persons with continuous complex care needs. J Am Geriatr Soc. 2003 Apr;51(4):549-55. doi: 10.1046/j.1532-5415.2003.51185.x. PMID 12657078